CLINICAL TRIAL: NCT01579682
Title: Adaptive Family Treatment for Adolescent Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, James Dale Lock, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPO 49694; SPO 49798 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2012-04-05; First posted 2012-04-18 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Anorexia Nervosa
Keywords: Eating Disorder; Anorexia Nervosa; Eating Disorder Not Otherwise Specified; Maudsley; Family-Based Therapy; FBT; Family Therapy
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychotherapy (Experimental): Family-Based Therapy (12 sessions)
  Interventions: Behavioral: Family-Based Therapy (FBT)
- Family-Based Therapy with Intensive Family-Focused Treatment (Experimental): The patient will receive 4 sessions of Family-Based therapy, and if the participant does not make adequate weight gain within this time period, will be assigned to Intensive Family-Focused Therapy (IFT).
  Interventions: Behavioral: Family-Based Therapy with Intensive Family-Focused treatment

INTERVENTIONS:
Behavioral: Family-Based Therapy (FBT) — 12 sessions of FBT over the course of 6 months.
  Arms: Psychotherapy
Behavioral: Family-Based Therapy with Intensive Family-Focused treatment — FBT for 4 weeks then Intensive Family-Focused treatment (IFT) should the participant not make adequate weight progress within the time frame.
  Arms: Family-Based Therapy with Intensive Family-Focused Treatment

SUMMARY:
Anorexia Nervosa (AN) has the highest mortality rate compared to any other psychiatric disorder. The most promising treatment for adolescents with AN is family-based treatment (FBT). However, only 50% of patients receiving FBT fully remit at 12-month follow-up. Consequently, providing an alternative therapy early in the treatment course for those not responding to FBT may enhance overall outcome. This study aims to develop a new treatment - Intensive Family-Focused Treatment (IFT) - to improve outcomes in those adolescents, aged 12-18 years, who do not show an early response to FBT.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for anorexia nervosa
* Lives with at least one English-speaking parent who is willing to participate
* Medically Stable
* Adequate transportation to clinic
* Proficient at speaking, reading, and writing English

Exclusion Criteria:

* Previous FBT for AN
* Medical condition that may affect eating or weight

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Full remission from AN (%MBW>95) | End of Treatment (6 months)
  Weight restoration to at least 95% of Median body weight (calculated by height, weight, gender, and age)

SECONDARY OUTCOMES:
Changes in subscale scores of the EDE | End of Treatment (6 months)
  Eating Disorder Examination subscale measures (weight concern, shape concern, dietary restraint) within 1 standard deviation of normative scores.

CONTACTS AND LOCATIONS:
Overall Officials: James D Lock, MD, PhD, Principal Investigator — Stanford University; Daniel LeGrange, PhD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Chicago, Chicago, Illinois

REFERENCES:
- See also: Related information — http://edresearch.stanford.edu